CLINICAL TRIAL: NCT01460875
Title: Pilot Study of IFN-alpha-2b Dose Reduction With Dose Optimization
Brief Title: Recombinant Interferon Alfa-2b in Treating Patients With Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Carson (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor-Investigator, William Carson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-07033; NCI-2011-03121 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT00634127 (obsolete NCT alias)
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Stage IA Skin Melanoma; Stage IB Skin Melanoma; Stage IIA Skin Melanoma; Stage IIB Skin Melanoma; Stage IIC Skin Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
Keywords: high risk melanoma; lymph node disease
MeSH Terms: conditions — Melanoma | interventions — Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (interferon therapy) (Experimental): Patients receive recombinant interferon alfa-2b SC thrice weekly. Treatment continues for 11 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: recombinant interferon alfa-2b; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: recombinant interferon alfa-2b — Given SC
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Intron A
Other: laboratory biomarker analysis — Blood for use in correlative studies approximately 30 ml 30 x 106 peripheral blood mononuclear cell (PBMCs) will be drawn on day 1 every other week during the first 12 weeks just prior to treatment and at 1 and 4 hours post therapy.
  Other Names: Correlative studies

SUMMARY:
This pilot clinical trial studies recombinant interferon alfa-2b in treating patients with melanoma. Recombinant interferon alfa-2b may interfere with the growth of tumor cells and slow the growth of melanoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether selection of the optimal IFN-alpha-2b (recombinant interferon alfa-2b) dose can be made using signal transduction data.

SECONDARY OBJECTIVES:

I. To determine the tolerability of adjuvant IFN-alpha-2b administered at an optimized dose in terms of the toxicities that are observed and the ability of patients to receive a full year of therapy.

II. The transcription of a panel of IFN-alpha-induced genes previously identified by microarray analysis will be determined by Real-Time reverse transcriptase-polymerase chain reaction (RT PCR) in order that the correlation between signal transducer and activator of transcription 1 (STAT1) phosphorylation and IFN-alpha gene regulation can be evaluated.

III. Microarray analysis of patient peripheral blood mononuclear cells (PBMCs) will be used to evaluate the effect of dose-reduction on IFN-alpha gene expression.

IV. In order to define the clinical role of tumor sensitivity to IFN-alpha, patient tumor biopsies taken prior to the administration of IFN-alpha will be systematically evaluated for cellular levels of janus kinase (Jak)-STAT signaling intermediates.

OUTLINE:

Patients receive recombinant interferon alfa-2b subcutaneously (SC) thrice weekly. Treatment continues for 11 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be considered a candidate for adjuvant IFN-alpha-2b therapy after having undergone successful surgery for high-risk melanoma (Breslow thickness > 4 mm or lymph node disease) or complete resection of metastatic disease; definitive surgery should have been accomplished no greater than 90 days prior to start of treatment with intravenous IFN-alpha-2b
* Patients must have completed 20 treatments of intravenous IFN-alpha-2b according to standard practice within 2 months of beginning treatment on this study
* Patients must have not have any evidence of persistent or recurrent disease as determined by the appropriate radiologic imaging techniques
* Patients may have received prior IFN-alpha therapy for metastatic disease, but more than 6 months must have passed between the last dose of IFN-alpha therapy for metastatic disease and the first dose of intravenous IFN-alpha-2b; patients who have had prior interleukin (IL)-2 are eligible for this study
* Patients may have received radiation therapy after intravenous IFN-alpha-2b; they may begin subcutaneous dosing of IFN-alpha-2b on this study after the radiation therapy has been completed; the patient may initiate dose reductions after the last radiation treatment as long as the appropriate amount of time has passed
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 70%)
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin =< 2.0 (Gilbert's disease permitted)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) < 3 x institutional upper limit of normal
* Creatinine =< 1.5 and stable OR
* Creatinine clearance >= 60 mL.min/1.73 m^2 for patients with creatinine levels above normal
* Pulse oximetry >= 90% on room air at rest
* Serum pregnancy test negative
* The effects of interferon alpha-2b on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, and because interferons are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* All patients must be informed of the investigational nature of this study and must provide written informed consent in accordance with institutional and federal guidelines; a copy of the informed consent document signed by the patient must be given to the patient

Exclusion Criteria:

* Patients may not be receiving any investigational agents
* History of allergic reactions attributed to compounds that are similar to interferon alpha-2b
* Patients known to be positive for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbsAg) or hepatitis C antibody
* Patients with organ allografts or immunodeficiency syndromes
* Patients with prior malignancies may participate provided they have been free of disease for at least 2 years except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; a history of depression in and of itself is not an exclusion to going participating provided the patient and physician believe the depression is controlled and the patient will discontinue the IFN-alpha should symptoms recur
* Pregnant women are excluded from this study because interferon alpha-2b is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IFN-alpha, breastfeeding should be discontinued if the mother is treated with IFN-alpha
* Prisoners will be excluded due to the need for multiple timed visits

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-04-22 (Actual); Primary Completion 2014-01-05 (Actual); Study Completion 2014-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer@osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Interferon Therapy)
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 52 [22 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Level of Activated STAT1(Phospho-STAT1)
Description: Mean and 95% confidence interval will be summarized for phospho-STAT1 at a lower dose and the standard dose. The phospho-STAT1 will also be compared between the dose levels.
Time Frame: up to 4 weeks
Measure: Mean (95% Confidence Interval); unit: MU/m2
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 34
MU/m2
  Dose I (10 MU/m2) | 5.96 [0.31 to 19.1]
  Dose II (4 MU/m2) | 4.80 [0.11 to 21.17]
Statistical Analysis 1: Comparison: Treatment (Interferon Therapy); Test type: Non-Inferiority — The method to be developed will allow us to declare that a response at a lower dose is not inferior to that at the standard dose for a particular patient, using a patient specific inferiority test; p = .22, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Patients With Adverse Events
Description: Determine the tolerability of adjuvant IFN-α-2b administered at an optimized dose in terms of the toxicities that are observed and the ability of patients to receive a full year of therapy.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 34
Participants | 15

3. Secondary Outcome: Percentage of Patients With Correlation Between STAT1 Phosphorylation and Interferon Alfa Gene Regulation
Description: Levels of p-STAT1 in PBMCs were analyzed just prior to IFN-a-2b administration to determine levels that remained stable or increased over the course of dose reduction.
Time Frame: Prior to treatment and 1 and 4 hours post therapy on day 1 every other week during the first 12 weeks, and then every 3 months
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 34
percentage of patients | 71

4. Secondary Outcome: Effect of Dose-reduction on Expression of Interferon Alfa Stimulated Genes
Description: Evaluated using microarray analysis of patient PBMCs. Compared using the Wilcoxon signed rank test for the dose 10MU/m2
Time Frame: 1 hour post therapy
Measure: Median (Full Range); unit: fold change
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 23
fold change
  SOCS1-1 hour post 10MU- | 1.5 [0.6 to 6.2]
  OAS1-1 hour post 10MU- | 1.6 [0.5 to 24.8]
  CXCL10-1 hour post 10MU | 28.7 [0.2 to 5128.0]
  CD69-1 hour post 10MU | 1.3 [0.4 to 12.1]

5. Secondary Outcome: Effect of Dose-reduction on Interferon Alfa Gene Expression
Description: Evaluated using microarray analysis of patient PBMCs. Compared using the Wilcoxon signed rank test for the dose 4MU/m2
Time Frame: 1 hour post therapy
Measure: Median (Full Range); unit: fold increase
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 23
fold increase
  SOCS1-1 hour post 4MU | 1.2 [0.4 to 17.7]
  OAS1-1 hour post 4MU | 1.6 [0.5 to 5.1]
  CXCL10-1 hour post 4MU | 6.0 [0.0 to 386.4]
  CD69-1 hour post 4MU | 1.3 [0.4 to 2.1]

6. Secondary Outcome: Effect of Dose-reduction on Interferon Alfa Gene Expression Through Marker CD69
Description: Evaluated using microarray analysis of patient PBMCs. Compared between doses using the Wilcoxon signed rank test.
Time Frame: 4 hours post therapy
Measure: Median (Full Range); unit: fold increase
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 22
fold increase
  SOCS1- 4 hour post-10MU | 1.5 [0.6 to 6.2]
  OAS1-4 hour post -10MU | 1.6 [0.5 to 24.8]
  CXCL10-4 hour post- 10MU | 28.7 [0.2 to 5128.0]
  CD69-4 hour post- 10MU | 1.3 [0.4 to 12.1]

7. Secondary Outcome: Effect of Dose-reduction on Interferon Alfa Gene Expression at Dose Level 4MU
Description: Evaluated using microarray analysis of patient PBMCs. Compared between doses using the Wilcoxon signed rank test.
Time Frame: 4 hours post therapy
Measure: Median (Full Range); unit: fold increase
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 23
fold increase
  SOCS1-4 hour post 4MU- | 1.6 [0.4 to 8.8]
  OAS1-4 hour post 4MU | 3.9 [0.4 to 19.1]
  CXCL10-4 hour post 4MU | 112.9 [0.0 to 2898.0]
  CD69-4 hour post 4MU | 1.5 [0.4 to 4.5]

8. Secondary Outcome: Clinical Role of Tumor Sensitivity to Recombinant Interferon Alfa-2b Using Cellular Levels of Jak-STAT Signaling Intermediates
Description: Define the clinical role of tumor sensitivity to IFN-α, patient tumor biopsies taken prior to the administration of IFN-α will be systematically evaluated for cellular levels of Jak-STAT signaling intermediates.
Time Frame: Baseline and every other week prior to recombinant interferon alfa-2b administration
Population: Data was not collected and analyzed for outcome measure
Arm/Group | Treatment (Interferon Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Interferon Therapy)
Serious Adverse Events (participants affected / at risk) | 22/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Interferon Therapy) (N=34)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Myelosuppression (Blood and lymphatic system disorders) | 7 (7)
Increased AST (Investigations) | 2 (2)
Neuropsychiatric Systems (Psychiatric disorders) | 2 (2)
Electrolyte Abnormalities (Metabolism and nutrition disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Interferon Therapy) (N=34)
Fever (General disorders) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (28)
Nausea (Gastrointestinal disorders) | 16 (16)
Vomiting (Gastrointestinal disorders) | 8 (8)
Fatigue (General disorders) | 28 (28)
Mylosuppression (Blood and lymphatic system disorders) | 27 (27)
Increased AST (Investigations) | 19 (19)
Neuropsychiatric Symptoms (Psychiatric disorders) | 12 (12) — including depression
Rigors/Chills (General disorders) | 19 (19)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Electrolyte Abnormalities (Metabolism and nutrition disorders) | 23 (23)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes